CLINICAL TRIAL: NCT07039006
Title: Error Augmentation for Upper Limb Rehabilitation in Stroke Survivors: a Proof-of-concept Study
Brief Title: Error Augmentation for Upper Limb Rehabilitation in Stroke Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Mindy F. Levin, Professor Mindy F. Levin, McGill University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MP-50-2020-1209
Record Dates: First submitted 2025-06-09; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Stroke
Keywords: stroke; motor learning; error augmentation; reaching
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training with EA feedback (Experimental): Subjects will undergo reaching training that includes EA feedback as a 30-degree elbow flexion error.
  Interventions: Behavioral: Training with EA feedback
- Training without EA feedback (Sham Comparator): Subjects will undergo reaching training that does not include EA feedback.
  Interventions: Behavioral: Training without EA feedback

INTERVENTIONS:
Behavioral: Training with EA feedback — Subjects will undergo reaching training that includes a 30-degree elbow flexion error 3 times in 1 week.
  Arms: Training with EA feedback
Behavioral: Training without EA feedback — Subjects will undergo reaching training that does not include EA feedback 3 times in 1 week.
  Arms: Training without EA feedback

SUMMARY:
Stroke can severely limit a person's ability to move their arm, especially when trying to reach by extending the elbow. These challenges often persist long after the stroke and make everyday activities more difficult. The investigators are testing a feedback strategy called error augmentation (EA) feedback that intentionally exaggerates movement errors to promote motor learning.

In this study, the investigators designed a virtual reality training program that uses EA feedback to encourage people with chronic stroke to use more elbow extension during reaching. The EA feedback makes it appear as though the elbow is more bent than it actually is, prompting the participant to extend their elbow further than they normally would. By having the patient practice movement with enhanced feedback, the investigators predict that the patient will increase the range of motion and improve reaching ability.

This is a short, proof-of-concept study to evaluate whether EA feedback shows early promise for improving arm movement in people with upper limb motor impairment after stroke. Participants are randomly assigned to either an EA training group or a control group (no-EA feedback). Each person completes three 30-minute virtual reality training sessions over 1 week. The investigators assess arm movement and motor impairment before and after training, and again one hour after the training to determine if improvements are retained.

Findings from this preliminary study will help determine whether this EA-based training approach should be used in a longer 9-week clinical trial aimed at promoting long-term recovery of arm function after stroke.

ELIGIBILITY:
Inclusion Criteria:

* Sustained a first-ever cortical/sub-cortical ischemic/hemorrhagic stroke ≥6 mo and ≤5 yr previously
* Has no medical complications
* Has arm paresis but can voluntarily flex/extend the elbow ~30 degrees
* Can provide informed consent

Exclusion Criteria:

* Has other major neurological or musculoskeletal problems that would interfere with task performance
* Has marked elbow proprioceptive deficits (<6/12 Fugl-Meyer Assessment for the Upper-Limb (FMA-UL) Sensation Scale)
* Has visuospatial neglect (Line Bisection Test)
* Has uncorrected vision
* Has depression (>14 on Beck Depression Inventory II)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-05-29 (Actual); Study Completion 2025-05-29 (Actual)

PRIMARY OUTCOMES:
Change in whole arm active workspace area | Prior to training.
  The size of the active arm workspace area will be expressed as a ratio of the active workspace determined when the subject actively moves their arm through the horizontal workspace to the passive workspace that is defined by the examiner moving the arm through the same space.
Change in the trunk-based index of performance | Baseline, immediately post-training, 1 hour post intervention.
  Described as a measure of reaching precision accounting for accuracy and speed of reaching together with the amount of trunk compensation.
Change in elbow extension angle at reaching offset | Baseline, immediately post-training, 1 hour post intervention.
  Elbow extension during a functional Test Task is calculated based on vectors between the markers placed on the acromion and the lateral epicondyle and between the lateral epicondyle and ulnar head of the affected arm. Arm movement onset/offset will be determined as the times at which the velocity of the endpoint marker increases/decreases and remains above/below 10% of the peak velocity.

SECONDARY OUTCOMES:
Change in endpoint accuracy | Baseline, immediately post-training, 1 hour post intervention.
  The x,y root mean square distance between the endpoint marker and the target at the end of a reaching movement.
Change in movement time | Baseline, immediately post-training, 1 hour post intervention.
  The time between the onset and offset of the movement.
Change in path smoothness | Baseline, immediately post-training, 1 hour post intervention.
  The number of peaks on a tangential velocity trace of each reaching trial.
Change in path straightness | Baseline, immediately post-training, 1 hour post intervention.
  Described using the index of curvature where the ratio between the actual movement path and a straight line path between the initial and final targets.

CONTACTS AND LOCATIONS:
Overall Officials: Mindy F Levin, PT, PhD, Principal Investigator — School of Physical and Occupational Therapy, McGill University
Locations (1):
- Jewish Rehabilitation Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
Data will be used for the purposes of this study only.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-05): https://cdn.clinicaltrials.gov/large-docs/06/NCT07039006/Prot_SAP_000.pdf
  • Informed Consent Form (2021-02-05): https://cdn.clinicaltrials.gov/large-docs/06/NCT07039006/ICF_001.pdf